CLINICAL TRIAL: NCT03147521
Title: Stepped Wedge Cluster Randomized Controlled Trial for the Evaluation of Effectiveness of a Accidental Falls Care Bundle Implementation in Elderly Hospital Patients.
Brief Title: Accidental Falls Care Bundle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Daniela Mosci, Registered Nurse, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 76/2014/O/Sper
Record Dates: First submitted 2017-05-04; First posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Accidental Falls
MeSH Terms: interventions — Patient Care Bundles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accidental falls care bundle (Experimental): Care Bundle Implementation Arm
  Interventions: Other: Care bundle
- Accidental falls standard care (Active Comparator): Standard Care Implementation Arm (Universal strategy application for the environmental and patient)
  Interventions: Other: Care bundle

INTERVENTIONS:
Other: Care bundle — Risk fall assessment at hospital admission with Conley scale or with findings of specific risk characteristics (previous falls, cognitive impairment, neuropsychological damage, increased need to go to the bathroom for increased evacuative needs, neuroleptic or cardiovascular drugs assumption); if risk is found shear the information with the team, writing it in patient chart, and positioning a specific symbol on patient bed. Inform patient and family about fall risk and ask, if possible, a continuous caregiver presence. Universal strategy application for the environmental safety and patient safety. Periodic assessment of drugs therapy, with the aim of reduce those that acts on central nervous system and cardiovascular system. If patient is at risk and alone, verify each 2 hours the need to go to the bathroom, change position or drink.

SUMMARY:
Accidental falls represents an elderly very important health problem, both in the community and within the hospital. The aim of this research project is to evaluate the effectiveness of accidental falls prevention care bundle in geriatrics, internal medicine, post acute, and rehabilitation wards, in terms of incidence and outcome reduction. It will be also investigated the cost effectiveness ratio, in terms of falls avoided, care bundle implementation costs, and falls related healthcare costs. The study will permit to evaluate the implementation feasibleness in time, considering the study will last for 20 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ≥ 75 years of age with or without documented fall risk and patients with < 75 years of age, but ≥ 18, only at documented fall risk, admitted at participant wards. The risk assessment will be performed with Conley scale and/or on the base of some specific fall risk characteristics (previous falls, cognitive impairment, neuropsychological damage, increased need to go to the bathroom for increased evacuative needs, neuroleptic or cardiovascular drugs assumption);
* Patients (or legal guardian for those incapable of giving their consent) that give their consent to the study participation .

Exclusion Criteria:

* Patients or legal guardian that don't give their consent to study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2016-12-28 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Falls Incidence rate | 5 months
  Number of accidental falls respect number of hospital days of stay in elderly hospital patients at the end of a 5 months step.

SECONDARY OUTCOMES:
Falls outcome | 5 monts
  Numbers falls from wich a fractures or a brain haemorrhage has been generated
Cost-effectiveness | 20 months
  Cost effectiveness ratio in terms of costs and avoided falls. Cost Implementation costs: costs for education and staff meeting; printed material costs.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Di Gennaro G, Chamitava L, Pertile P, Ambrosi E, Mosci D, Fila A, Alemayohu MA, Cazzoletti L, Tardivo S, Zanolin ME. A stepped-wedge randomised controlled trial to assess efficacy and cost-effectiveness of a care-bundle to prevent falls in older hospitalised patients. Age Ageing. 2024 Jan 2;53(1):afad244. doi: 10.1093/ageing/afad244. PMID 38251740